CLINICAL TRIAL: NCT05756218
Title: The Effect of Taboo Game Adapted for Nursing Diagnoses in Professional Practice Lesson on Motivation and Perception of Nursing Diagnoses in Nursing Students: A Randomized Controlled Study
Brief Title: Motivation of Nursing Students and Perception Levels of the Taboo Game Adapted for Nursing Diagnoses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Tuba KORKMAZ ASLAN, Asist. Prof. Tuba KORKMAZ ASLAN Ph.D., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Taboo Game Nursing Diagnoses
Record Dates: First submitted 2023-01-25; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Nursing Diagnosis; Taboo Game; Motivation
Keywords: Nursing Diagnosis Perception; Taboo Game; Motivation

STUDY DESIGN:
Intervention Model Description: It was designed as a parallel group randomized controlled trial. The reporting of the study was planned in accordance with the PEER criteria
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding; groups 'X" and "Y" are named as independent statistical posts statistical blinding, blinding the educational staff conducting the professional practice course, blinding the person preparing the randomization table and the control group. In order for the control group to be blinded, this group was planned from another faculty.
  Randomization below will be performed by a statistical specialist other than randomization researchers for the purpose of preventing bias and ensuring confidentiality. He will not know which of the lecturers who are lecturing in both groups are in the experimental group and who are in the control group. Statistical analyzes were performed and after the research report is written, the encodings made for the intervention and control group will be opened. Blinding will be provided in terms of collecting and reporting departmental research data. By an independent statistic in random ranking list order random.org made on site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Obtaining Consent, Demographic Information Form, Teaching Material Motivation Scale and Nursing Diagnosis Perception Scale face-to-face filling Playing the game with nursing diagnosis taboo cards prepared on the day of no practice for 7 weeks
  Interventions: Other: nursing diagnoses - taboo game
- Control (No Intervention): Obtaining Consent, Demographic Information Form, Teaching Material Motivation Scale and Nursing Diagnosis Perception Scale face-to-face filling Continuing the application as in the curriculum for 7 weeks

INTERVENTIONS:
Other: nursing diagnoses - taboo game — Playing 7 weeks nursing diagnoses taboo cards
  Arms: Experiment

SUMMARY:
The goal of this To determine the effect of the taboo game adapted for nursing diagnoses in the professional practice course on the motivation and perception levels of nursing diagnoses in nursing students.

Type of Research:

It was designed as a parallel group randomized controlled trial. The reporting of the study was planned in accordance with the PEER criteria] in [describe participant population/health conditions]. The main question[s] it aims to answer are:The Research Hypothesis: H1: The taboo game organized for nursing diagnoses in the professional practice course has an effect on the motivation of nursing students.

H2: The taboo game organized for nursing diagnoses in the professional practice course has an effect on nursing students' perception of nursing diagnoses.

Participants will [The Universe of her Research: The universe of her research Necmettin Erbakan University Faculty of Nursing 4. Class (Quota: 145) and Necmettin Erbakan University Seydişehir Kamil Akkanat SBF Nursing department 4. The class (Quota: 42) students will be formed].

If there is a comparison group: It was increased by 10% for possible records, the research was planned to be completed with 80 people, with an error of 0.05, a power of 0.80 and an effect size of 0.600; 40 experiments, 40 control groups.

DETAILED DESCRIPTION:
The other measure to be used in the study is the scale of perception of nursing definitions. In this calculation, the results of a study that looked at the perception of citizenship definitions of students were used. In the study in question, the scores of student nurses' choice of profession (101.95±18.29) and choice of profession (98.53±16.57) perception of citizenship definitions are different (Su & Kose 2021). In the study, SDSpooled was calculated because the number of people in the groups was not equal (n1: 203, n2=79). The formula √ [(n1-1)212+(n2-1)222]/n1+n2-k was used in the calculation (SDpooled= 0.35). The results obtained were calculated in the G*Power3.1.9.4 package program. According to this calculation, the number of people to be reached with 0.05 error, 0.80 power and 0.600 effect size was determined as 36 people as the experimental group, 36 people as the control group, and a total of 72 students for the control and experimental group. It was increased by 10% for possible records, the research was planned to be completed with 80 people, with an error of 0.05, a power of 0.80 and an effect size of 0.600; 40 experiments, 40 control groups.

Randomization and Blinding:

Experimental group Necmettin Erbakan University Seydişehir Kamil Akkanat SBF Nursing department 4. Class students, control group Necmettin Erbakan University Faculty of Nursing 4. Class students will be formed. The class lists will be used depending on the list order taken from the school. Random.org according to the randomization table made from , the assignment will be made from their list. The experimental group "X" will be called the control group "Y".

Blinding; groups 'X" and "Y" are named as independent statistical posts statistical blinding, blinding the educational staff conducting the professional practice course, blinding the person preparing the randomization table and the control group. In order for the control group to be blinded, this group was planned from another faculty. The experimental group and the researchers were not blinded.

Randomization below will be performed by a statistical specialist other than randomization researchers for the purpose of preventing bias and ensuring confidentiality. He will not know which of the lecturers who are lecturing in both groups are in the experimental group and who are in the control group. Statistical analyzes were performed and after the research report is written, the encodings made for the intervention and control group will be opened. Blinding will be provided in terms of collecting and reporting departmental research data. By an independent statistic in random ranking list order random.org made on site.

Data Collection Techniques and Tools: The taboo game has been adapted to meet the content and organization of the professional practice course, which is 27 ECTS (32 Applications) compulsory for fourth grade students in the spring semester. The goal of the game is for the individual to make his partner guess as many primary (WIP) words as possible in a given time, without using the "taboo" words to describe the main term. The one who correctly defines the most basic words wins. The creation of playing cards is as follows; the cards will be prepared using nursing diagnostics. At Taboo (Hasbro Inc., Pawtucket, RI), a person is given a set of cards containing both the primary word or phrase and five "taboo" words. The primary word (WIP) at the top of each card is clearly separated from the five taboo words at the bottom. For example, the taboo words under the WIP "constipation" may be "rectum", "great ablution", "diarrhea", "buttocks" and "excretion". Taboo words can be adjusted according to the student's level and difficulty, and the cards can be laminated for repeated use. Finally, a voice alert and a 1-minute timer (eg. October Jul. Additional materials will be provided, including (hourglass) (Lofton 2022).

NANDA Nursing diagnoses are grouped according to functional health patterns and according to this distribution; Health perception-Health Management 10 cards, Nutritional-Metabolic card 15, excretory, 15 cards and gas exchange, Activity/rest for 25 cards, perception/Cognition 8 cards, self-image 6 Cards, Role-relationship 10 cards, 4 cards, Sexuality, coping/stress tolerance, 30 Card, 6 card Life Principles, safety/protection card 30, the comfort, the card 8, and growth/Development, so it will be 3 cards in total, 170 card will be issued.

The students of the experimental group will be asked to follow the following rules by playing the taboo game created with that topic every week after the lesson:

1. A person from the research team comes with a set of playing cards in his hand and starts the game.
2. Students have one minute to guess as many terms as possible.
3. Another person who is on the research team is next to the student to make sure that he does not use the words "taboo" and to save time.
4. A student cannot skip terms right away when defining words. If the student is experiencing a certain difficulty, someone from the team can help. The student can move to the next one only after the allotted time (∼ 10-15 seconds).

Below are the NANDA Nursing diagnoses grouped according to functional health patterns:

1. Health Promotion
2. Nutrition
3. Discharge and Gas Exchange
4. Activity/Recreation
5. Perception/Cognition
6. Self-Perception
7. Role relationship
8. Sexuality
9. Coping/Stress tolerance
10. Life principles
11. Security/Protection
12. Comfort
13. Growth/Development Both the control group (Konya-Nursing 4. Class) as well as students in the experimental group (Seydişehir-Nursing 4. Class) takes the internship application course with the same credit. The application is carried out in the same hospital. Similar programs are implemented in both schools.

Before the taboo game, obtaining Consent, Demographic information form, Teaching Materials Motivation Scale and Nursing Diagnosis Perception Scale will be applied to both groups. Together with the experimental group, the taboo game prepared for two of the groups according to the functional health patterns of NANDA Nursing diagnoses will be played every week. The cards prepared about the subject are written next to each subject. after the 7-week period is over, the Teaching Materials Motivation Scale and the Nursing Diagnosis Perception Scale will be applied again.

Data Collection: After the data of the research are approved by the Ethics Committee and the permissions of the institution are obtained, the first data will be collected on February 06, 2023 and the taboo game will start to be played. It is planned to collect the latest data on March 25, 2023. The data will be collected by filling in face-to-face by the researchers. Nursing diagnoses taboo game will be played for a total of 7 weeks on the day when students who practice 4 days every week do not practice.

Variables of the Research Dependent variables; Teaching Materials Motivation Scale total score and Nursing Diagnosis Perception Scale total score Independent variables; sociodemographic characteristics and taboo game application

ELIGIBILITY:
Inclusion Criteria:

1. NEU Faculty of Nursing 4. Becoming a classroom teacher
2. NEU Seydişehir Kamil Akkanat SBF Nursing Department 4. Becoming a classroom teacher
3. To be taking the Profession Application course for the first time
4. to indicate that he will be eligible to actively participate in the taboo game at the end of 7 weeks
5. Willingness to participate in the study of their own free will (representative informed consent)

Exclusion Criteria:

1) He does not understand Turkish, does not read and does not understand

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-27 (Estimated); Primary Completion 2023-03-24 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
Time Frame | 1 day
  a day before the taboo game Obtaining Consent, Demographic Information Form, to measure motivation Teaching Material Motivation Scale face-to-face filling
  Sociodemographic Information Form: The literature was reviewed and prepared by the researchers. The form consists of 9 questions in total.
  Teaching Materials Motivation Scale: It is a 24-item scale. This scale consists of two sub-dimensions: "attention-attention" and "confidence-satisfaction". The lowest score that can be obtained from the scale is 24, and the highest score is 120.
Time Frame | 1 day
  a day before the taboo game, to measure the perception levels of nursing diagnoses Nursing Diagnosis Perception Scale face-to-face filling The Nursing Diagnosis Perception Scale: Scale consists of 26 items in total. The total scale score ranges from 1 to 5. Dec. The low total score obtained from the scale shows that nurses perceive nursing diagnoses in a positive way. The subfields of the scale are also calculated as the total score of the scale.

SECONDARY OUTCOMES:
Time Frame | 7 weeks
  at the time end of 7 weeks, to measure motivation Teaching Material Motivation Scale face-to-face filling
  Sociodemographic Information Form: The literature was reviewed and prepared by the researchers. The form consists of 9 questions in total.
  Teaching Materials Motivation Scale: It is a 24-item scale. This scale consists of two sub-dimensions: "attention-attention" and "confidence-satisfaction". The lowest score that can be obtained from the scale is 24, and the highest score is 120.
Time Frame | 7 weeks
  at the time end of 7 weeks, to measure the perception levels of nursing diagnoses Nursing Diagnosis Perception Scale face-to-face filling
  The Nursing Diagnosis Perception Scale: Scale consists of 26 items in total. The total scale score ranges from 1 to 5. Dec. The low total score obtained from the scale shows that nurses perceive nursing diagnoses in a positive way. The subfields of the scale are also calculated as the total score of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Türkben Polat, PhD, Study Chair — hturkbenpolat@erbakan.edu.tr

REFERENCES:
- [Background] Boctor L. Active-learning strategies: the use of a game to reinforce learning in nursing education. A case study. Nurse Educ Pract. 2013 Mar;13(2):96-100. doi: 10.1016/j.nepr.2012.07.010. Epub 2012 Aug 19. PMID 22910398
- [Background] Karaca T, Aslan S. Effect of 'nursing terminologies and classifications' course on nursing students' perception of nursing diagnosis. Nurse Educ Today. 2018 Aug;67:114-117. doi: 10.1016/j.nedt.2018.05.011. Epub 2018 May 23. PMID 29857304
- [Background] Kim SC, Jillapali R, Boyd S. Impacts of peer tutoring on academic performance of first-year baccalaureate nursing students: A quasi-experimental study. Nurse Educ Today. 2021 Jan;96:104658. doi: 10.1016/j.nedt.2020.104658. Epub 2020 Nov 7. PMID 33186748
- [Background] Lofton CM. Laying the Foundation for Critical Thinking With the Nursing Taboo Game. J Nurs Educ. 2022 Jun;61(6):355. doi: 10.3928/01484834-20220404-05. Epub 2022 Jun 1. No abstract available. PMID 35667116
- [Background] Mousavinasab ES, Rostam Niakan Kalhori S, Zarifsanaiey N, Rakhshan M, Ghazisaeedi M. Nursing process education: A review of methods and characteristics. Nurse Educ Pract. 2020 Oct;48:102886. doi: 10.1016/j.nepr.2020.102886. Epub 2020 Sep 15. PMID 32961511
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Pitkanen S, Kaariainen M, Oikarainen A, Tuomikoski AM, Elo S, Ruotsalainen H, Saarikoski M, Karsamanoja T, Mikkonen K. Healthcare students' evaluation of the clinical learning environment and supervision - a cross-sectional study. Nurse Educ Today. 2018 Mar;62:143-149. doi: 10.1016/j.nedt.2018.01.005. Epub 2018 Jan 30. PMID 29353088
- [Background] Sanson G, Vellone E, Kangasniemi M, Alvaro R, D'Agostino F. Impact of nursing diagnoses on patient and organisational outcomes: a systematic literature review. J Clin Nurs. 2017 Dec;26(23-24):3764-3783. doi: 10.1111/jocn.13717. Epub 2017 Feb 23. PMID 28042921
- [Background] Yu M, Tong H, Li S, Wu XV, Hong J, Wang W. Clinical competence and its association with self-efficacy and clinical learning environments among Chinese undergraduate nursing students. Nurse Educ Pract. 2021 May;53:103055. doi: 10.1016/j.nepr.2021.103055. Epub 2021 Apr 16. PMID 33951599